CLINICAL TRIAL: NCT07284953
Title: A Pilot, Single Arm Post-Market Clinical Study to Demonstrate the Feasibility, Safety and Efficacy of PuraBond™ Absorbable Haemostatic Material for the Management of Bleeding and Tissue Healing in Robotic Partial Nephrectomy
Brief Title: A Novel Haemostatic Agent for Robotic Partial Nephrectomy
Acronym: PuraBond
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024SUR137
Record Dates: First submitted 2025-11-14; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Kidney Cancer; Renal Cell Carcinoma
Keywords: Robotic Partial Nephrectomy; PuraBond
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to PuraBond or standard care of Floseal to stop the bleeding after renorrhaphy suture when undergoing a robotic partial nephrectomy procedure (primary resection).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PuraBond (Experimental): Collect medical information on patients who were treated with PuraBond during robotic partial nephrectomy, according to each participating institution's procedures and standards of care.
  Evaluate the feasibility, safety and efficacy of PuraBond in achieving haemostasis and post operative healing at the resection site compared to standard of care agent for robotic partial nephrectomy procedures
  Interventions: Device: PuraBond

INTERVENTIONS:
Device: PuraBond — Consecutive patients undergoing robotic partial nephrectomy procedure (primary resection) and treated with PuraBond

SUMMARY:
Kidney cancer is one of only a few cancers with an increasing incidence over the past two decades. Renal cell carcinoma (RCC) accounts for over 85% of all kidney tumours, which makes up 2-3% of all adult malignancies. Approximately, 70% of RCCs are incidentally discovered on axial imaging of the abdomen with >50% of RCCs being low-stage (T1-T2 N0M0). Despite advancements in drug discovery for advanced RCC, mortality rates have not changed over the past two decades, however for patients with the low-stage disease, surgical extirpation offers excellent 5-year survival rates of 95%.

Nephron-sparing surgery (NSS) provides effective curative therapy for patients with localized renal cell carcinoma with the benefit of kidney preservation and excellent cancer-specific survival. However, the most frequent complications during NSS, after tumour resection are bleeding, urinary fistula formation, and ischemic renal damage. More precisely, the urological complication was defined as significant haemorrhage >500 mL necessitating intervention or transfusion, urine leakage (drainage of greater than 50 mL daily for more than one week with fluid biochemistry compatible with urine) and acute renal failure (resulting in any dialysis, ureteral obstruction or kidney loss).

In the field of partial nephrectomy procedures, it is therefore crucial achieving adequate haemostasis intraoperatively during post tumour excision while the artery is clamped and after being unclamped.

DETAILED DESCRIPTION:
Kidney cancer is one of only a few cancers with an increasing incidence over the past two decades. Renal cell carcinoma (RCC) accounts for over 85% of all kidney tumours, which makes up 2-3% of all adult malignancies. Approximately, 70% of RCCs are incidentally discovered on axial imaging of the abdomen with >50% of RCCs being low-stage (T1-T2 N0M0). Despite advancements in drug discovery for advanced RCC, mortality rates have not changed over the past two decades, however for patients with the low-stage disease, surgical extirpation offers excellent 5-year survival rates of 95%.

Nephron-sparing surgery (NSS) provides effective curative therapy for patients with localized renal cell carcinoma with the benefit of kidney preservation and excellent cancer-specific survival. However, the most frequent complications during NSS, after tumour resection are bleeding, urinary fistula formation, and ischemic renal damage. More precisely, the urological complication was defined as significant haemorrhage >500 mL necessitating intervention or transfusion, urine leakage (drainage of greater than 50 mL daily for more than one week with fluid biochemistry compatible with urine) and acute renal failure (resulting in any dialysis, ureteral obstruction or kidney loss).

In the field of partial nephrectomy procedures, it is therefore crucial achieving adequate haemostasis intraoperatively during post tumour excision while the artery is clamped and after being unclamped.

Haemostatic agent can be used after Robotic-assisted laparoscopic partial nephrectomy (RLPN) or after the sutureless technique with bipolar cauterization of the surgical bed for the haemostatic control in the treatment of small cortical masses. It can be always used for tumours ≤1.5 cm and can be a valid option also for tumours between 1.6 and 2.5 cm, aside from their spatial extension.

As such, there is a need for the exploration of the use of novel haemostatic agents, such as self-assembling peptide (SAP)-based haemostat, to manage bleeding during partial nephrectomy.

The SAPs are oligopeptides (8 - 16 amino acids) composed of alternating hydrophilic and hydrophobic amino acids. These peptide chains can rapidly form nanofibers and create 3D microenvironments at a physiological pH and osmolarity. As peptides are nontoxic, biocompatible, and biodegradable, the SAPs can be used without an apparent immunological response, are also easy handling and are easy to inject due to their water solubility. Due to all these properties, SAPs are suitable for clinical use. One of the most widely studied SAPs is RADA16. It contains the amino acids alanine, lysine, and glutamate in repeated sequences of 4 X [Arg-Ala-Asp-Ala] (RADA16). RADA16 has proven utility as an effective topical haemostatic agent in a variety of surgical and pathological scenarios.

PuraStat and PuraBond (same product manufactured by 3-D Matrix Europe SAS, Caluire-et-Cuire, France) are CE-marked medical devices delivered by pre-filled syringes as viscous aqueous solutions of synthetic 2.5% RADA16. When RADA16 comes in to contact with blood or other physiological fluids, it forms a hydrogel. The hydrogel formation acts as a mechanical barrier and blocks the flow of the blood from the wound and thereby, demonstrates excellent topical haemostatic control. Initial preclinical studies investigating this peptide have shown other benefits in addition to its haemostatic properties, including improved wound healing.

Since 2014, PuraStat/PuraBond haemostatic efficacy has been significant successfully assessed in clinical studies, including in GI endoscopy, ENT, cardiovascular and general surgery (liver surgery) to support its use in humans demonstrated >90% of achieved haemostasis within 2min. There is a recent Australian case series published in Oct 2023 evaluating 29 patients undergoing nerve sparing robot-assisted radical prostatectomy, concluding it is a safe haemostatic agent.

However, there are no current studies published regarding self-assembling peptide haemostatic agents in partial nephrectomy. This study aims to generate clinical evidence investigating the feasibility and safety of PuraBond in achieving haemostasis in partial nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, aged 18 years or above
2. Patient has a clinical indication for laparoscopic partial nephrectomy procedure
3. Participant is willing and able to give informed consent for participation in the study
4. Intraoperative criteria: Subject requiring the use of PuraBond for persisting mild and moderate bleeding(s) when haemostasis by ligation or standard means are insufficient or impractical.

Exclusion Criteria:

1. Pregnant or Lactating women
2. Unable to give informed consent
3. Patient undergoing redo surgery
4. Fibrin glue and/or topical haemostatic agent used before or concomitantly to the use of PuraBond
5. Known allergy or hypersensitivity to any component of the investigational treatment PuraBond
6. Known coagulopathy
7. Clinical indication not satisfying inclusion criteria
8. Patient has clinical evidence of disease or condition expected to compromise survival or ability to complete follow-up assessments during the study duration
9. Patients currently participating in, or planning to enroll in another clinical study that may impact participation or outcomes of this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Intraoperative efficacy rate in stopping remaining mild and moderate bleeding after declamping within 2 minutes | During robotic partial nephrectomy procedure

SECONDARY OUTCOMES:
Time to Haemostasis after PuraBond application | During robotic partial nephrectomy procedure
The amount of PuraBond needed to achieve haemostasis | During robotic partial nephrectomy procedure
Ease of use of PuraBond (difficult or easy) | During robotic partial nephrectomy procedure
Rate of revision for bleeding | During robotic partial nephrectomy procedure
Radiomics score of tissue healing at 6 months post op CT scan | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No